CLINICAL TRIAL: NCT03548532
Title: Embryo Culture At a Constant Temperature of 36.6°C or 37.1°C: a Randomized Controlled Trial
Brief Title: Embryo Culture At a Constant Temperature of 36.6°C or 37.1°C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Neelke De Munck, PhD, Universitair Ziekenhuis Brussel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017/060
Record Dates: First submitted 2017-10-23; First posted 2018-06-07 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-01

CONDITIONS: Temperature; Extreme, Exposure
Keywords: temperature

STUDY DESIGN:
Intervention Model Description: Based on the randomisation list, patients fulfilling the inclusion criteria will be assigned to one of each arm. A total of 119 patients are needed in every arm in this superiority trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 36.6°C (Active Comparator): Embryos of these patients will be cultured at 36.6°C from day 0 after ICSI, untill day 6.
  Interventions: Device: G210 incubator
- 37.1°C (Experimental): Embryos of these patients will be cultured at 37.1°C from day 0 after ICSI, untill day 6.
  Interventions: Device: G210 incubator

INTERVENTIONS:
Device: G210 incubator — very stable culture temperature, up to 0.1°C, in both arms
  Other Names: Ksystems

SUMMARY:
On the day of oocyte retrieval, participants will be randomized to stable culture at 37.1°C or 36.6°C with the ultimate aim of finding a difference in clincial pregnancies.

DETAILED DESCRIPTION:
A previous study in our centre analysed stable embryo culture at 36.6°C and 37.1°C, on sibling oocytes. The primary aim was to analyse possible differneces in embryo development (utilization rate) up to day 5/6. In this study, the investigators found a high difference in clinical pregnancy rate between both groups (46.4% versus 77.4%). Since this study was not powered to find differences in clincial pregnancy rates between both groups, this RCT was especially powered as a superiority trial to find differences in clincial pregnancy rates between both groups. On the day of oocyte retrieval, patients will be allocated to culture at one of both temperatures.

ELIGIBILITY:
Inclusion Criteria:

* Day 5 transfer
* Single embryo transfer
* Only ejaculated sperm (fresh or frozen, autologous or heterologous)
* BMI <35
* Age <40 years
* Cycle rank <3 for the current child
* Last ultrasound: 8 follicles of at least 12 mm
* At least 6 mature oocytes

Exclusion Criteria:

* IVF
* IVF versus ICSI
* Failed fertilization in previous cycle
* no previous cycle without embryo transfer
* No use of Ca ionophores for embryo quality or fertilization problems

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 234 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2022-11-26 (Actual); Study Completion 2023-01-18 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy | 7 weeks
  ultrasound: sac and fetal heartbeat positive

SECONDARY OUTCOMES:
Fertilization rate | 1 day
  number of fertilized oocytes, per number of injected oocytes
embryo development/utilization rate | 6 days
  number of embryos transferred or cryopreserved per fertilized oocytes
live birth rate of the fresh cycle | 43 weeks
  number of live births per started cycle
cumulative live birth rate per cycle | 104 weeks
  fresh and frozen embryo transfer: outcome of the deliveries

CONTACTS AND LOCATIONS:
Overall Officials: Greta Verheyen, PhD, Study Director — UZBrussel
Locations (1):
- Universitair Ziekenhuis Brussel, Brussels, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: Yes
For statistical Analysis
Supporting Information: SAP
Time Frame: within 6 months after study completion
Access Criteria: Only relevant information will be given to the statistician (who is also a clinical doctor in our centre)
URL: http://www.brusselsivf.be

REFERENCES:
- [Derived] Wouters K, Mateizel I, Segers I, Van de Velde H, Van Landuyt L, De Vos A, Schoemans C, Jankovic D, Blockeel C, Drakopoulos P, Tournaye H, De Munck N. Clinical pregnancy rates after blastocyst culture at a stable temperature of 36.6 degrees C versus 37.1 degrees C: a prospective randomized controlled trial. Hum Reprod. 2024 Oct 1;39(10):2233-2239. doi: 10.1093/humrep/deae193. PMID 39241807